CLINICAL TRIAL: NCT04561505
Title: Holmium Laser Enucleation of the Prostate Versus Monopolar Transurethral Resection of the Prostate in Management of Benign Prostatic Hyperplasia.
Brief Title: HoLEP vs mTURP in Management of Benign Prostatic Hyperplasia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Salah Sayed, Dr., Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HoLEP
Record Dates: First submitted 2020-09-18; First posted 2020-09-23 (Actual); Last update posted 2020-09-23 (Actual); Status verified 2020-09

CONDITIONS: Prostatic Hyperplasia
Keywords: prostate; transurethral resection of prostate; HoLEP
MeSH Terms: conditions — Prostatic Hyperplasia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Holmium laser enucleation of prostate (Active Comparator): patients that undergo Holmium laser enucleation of prostate (HoLEP) procedure
  Interventions: Procedure: Holmium laser enucleation of prostate
- monopolar transurethral resection of prostate (Active Comparator): patients that undergo monopolar transurethral resection of prostate
  Interventions: Procedure: monopolar transurethral resection of prostate

INTERVENTIONS:
Procedure: Holmium laser enucleation of prostate — surgical management of BPH by Holmium laser enucleation using 0.9% saline fluid for irrigation
  Arms: Holmium laser enucleation of prostate
Procedure: monopolar transurethral resection of prostate — surgical management of BPH by monopolar TURP using distilled water for irrigation
  Arms: monopolar transurethral resection of prostate

SUMMARY:
To compare the clinical outcome regarding safety and efficacy between Holmium laser enucleation of the prostate and transurethral resection of the prostate in management of benign prostatic hyperplasia.

DETAILED DESCRIPTION:
Benign prostatic hyperplasia (BPH) affects 70% of men older than 70 years and is a significant cause of morbidity in this population.

The symptoms of BPH include impaired physiological and functional well-being, which interferes with daily living.

Lower urinary tract symptoms (LUTS) in elderly men are mainly related to an enlarged prostate, the actual link between an enlarged prostate and the onset of symptoms are multifactorial.

LUTS include both irritative symptoms in the form of urgency, frequency, nocturnal enuresis and urge incontinence as well as obstructive symptoms comprise hesitancy, weak interrupted stream of urine, incomplete voiding which eventually affect the quality of life (QoL), the main goal of treatment is resolve these symptom.

Multiple surgical options are available for management of benign prostatic hyperplasia (BPH) and its associated symptoms. Transurethral resection of the prostate (TURP) and open prostatectomy remain the gold standard surgical management. However, considerable morbidities are associated with both procedures and mainly related to the prostate size.

These complications may be either patient or surgically related. The patient's related complications are cardiac arrhythmia, myocardial infarction, pulmonary embolism, exacerbation of previous respiratory disease, deep venous thrombosis and death. The surgical related complication includes bleeding, capsular perforation, urosepsis, incontinence, conversion to open surgery, bladder neck stenosis, redo surgery and transurethral resection syndrome.

Clearly, a wide gap existed between simple medical therapy on one hand and TURP on the other hand. This wide gap is coupled with the need for a less morbid alternative to TURP that led to the emergence of various less invasive therapy among which Laser based minimally invasive procedure.

Modern laser therapy for BPH has advantages over TURP including decreased blood loss and minimal serum electrolyte changes resulting in fewer cardiovascular complications, decreased catheter time, shorter hospital stay and the ability to treat patients on anticoagulation.

Because of these potential advantages, there has been a shift in practice patterns with laser procedures accounting for 57% of surgical interventions for BPH, compared to traditional TURP which accounted for only 39% of interventions in 2005.

Holmium laser enucleation of the prostate (HoLEP) is the most recent step in the evolution of holmium laser prostatectomy. HoLEP is a safe and effective surgical procedure, which has comparable results to transurethral resection of the prostate (TURP) and open prostatectomy, with low morbidity and short hospital stay.

HoLEP is equally suitable for small, medium, and large prostate glands, with clinical outcomes that are independent of prostate size, and recently it has been proposed as a new gold standard for treatment of symptomatic benign prostatic hyperplasia (BPH). Currently, all BPH guidelines recommend HoLEP as a surgical treatment of BPH.

For a procedure to be considered a gold standard, it must provide effective results, low morbidity, and durable outcomes. HoLEP, as many of the new alternative treatments for symptomatic BPH, has scanty data regarding its role in Egyptian population and if it can replace TURP to be the gold standard.

To our best knowledge, no one estimated cost effectiveness between the two techniques in a developing country.

Our study aimed to compare the efficacy, safety and cost effectiveness of HoLEP versus monopolar TURP in management of benign prostatic hyperplasia in a developing country.

ELIGIBILITY:
Inclusion Criteria:

* prostate volume less than 80 ml
* high IPSS more than 19 affecting quality of life
* recurrent urinary retention with failure of medical treatment
* recurrent urinary tract infection
* affection of upper urinary tract
* refractory hematuria
* bladder stones
* bladder diverticula

Exclusion Criteria:

* patients with neurogenic bladder
* patients with previous prostate or urethral surgery
* associated urethral stricture
* prostate cancer diagnosed by TRUS biopsy
* prostate volume more than 80 ml

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — males only have prostate that will need surgical management of BPH
Enrollment: 60 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2020-02-01 (Actual); Study Completion 2020-02-29 (Actual)

PRIMARY OUTCOMES:
the international prostate symptom score (IPSS) | 1 year
  assessing the improvement of IPSS
maximum urine flow rate (Qmax) | 1 year
  assessing the improvement of Qmax

SECONDARY OUTCOMES:
operative time | immediately postoperative
  estimating the operative time in both groups in minutes
resected volume | immediately postoperative
  measuring the resected volume of prostate after each operation
postoperative drop in hemaoglobin level | 1 day postoperative
  comparing postoperative hemoglobin level with preoperative level in both groups
postoperative drop in sodium level | 1 day postoperative
  comparing postoperative sodium level with preoperative level in both groups
postoperative catheterization time | 4 days postoperative
  assessing postoperative catheterization time in both groups
duration of hospital stay | 3 days postoperative
  assessing duration of hospital stay in both groups
postvoiding residual urine volume | 1 year
  assessing postvoiding residual urine volume in both groups
ultrasound assessed prostate volume | 1 year
  comparing ultrasound assessed prostate volume in both groups

OTHER OUTCOMES:
cost analysis | 3 days postoperative
  comparing cost analysis for each patient in both groups as regards running cost including laser fiber or monopolar loop, irrigation fluid and cost of hospital stay.
complications | 1 year
  assessing intraoperative, early postoperative and late postoperative complications in both groups

CONTACTS AND LOCATIONS:
Overall Officials: Salah Sayed, master, Principal Investigator — assistant lecturer of urology, Ainshams university hospital, Cairo, Egypt; Amr Elshorbagy, PhD, Study Chair — professor of urology, Ainshams university hospital, Cairo, Egypt; Mahmoud A. Mahmoud, PhD, Study Chair — assistant professor of urology, Ainshams university hospital, Cairo, Egypt; Diaaeldin Mostafa, PhD, Study Director — assistant professor of urology, Ainshams university hospital, Cairo, Egypt
Locations (1):
- Ainshams university hospital, Cairo, Egypt

REFERENCES:
- [Background] Magoha GA. Medical management of benign prostatic hyperplasia: a review. East Afr Med J. 1996 Jul;73(7):453-6. PMID 8918007
- [Background] Oelke M, Bachmann A, Descazeaud A, Emberton M, Gravas S, Michel MC, N'dow J, Nordling J, de la Rosette JJ; European Association of Urology. EAU guidelines on the treatment and follow-up of non-neurogenic male lower urinary tract symptoms including benign prostatic obstruction. Eur Urol. 2013 Jul;64(1):118-40. doi: 10.1016/j.eururo.2013.03.004. Epub 2013 Mar 13. PMID 23541338
- [Background] Biester K, Skipka G, Jahn R, Buchberger B, Rohde V, Lange S. Systematic review of surgical treatments for benign prostatic hyperplasia and presentation of an approach to investigate therapeutic equivalence (non-inferiority). BJU Int. 2012 Mar;109(5):722-30. doi: 10.1111/j.1464-410X.2011.10512.x. Epub 2011 Aug 22. PMID 21883855
- [Background] Bach T, Muschter R, Sroka R, Gravas S, Skolarikos A, Herrmann TR, Bayer T, Knoll T, Abbou CC, Janetschek G, Bachmann A, Rassweiler JJ. Laser treatment of benign prostatic obstruction: basics and physical differences. Eur Urol. 2012 Feb;61(2):317-25. doi: 10.1016/j.eururo.2011.10.009. Epub 2011 Oct 21. PMID 22033173
- [Background] Rassweiler J, Teber D, Kuntz R, Hofmann R. Complications of transurethral resection of the prostate (TURP)--incidence, management, and prevention. Eur Urol. 2006 Nov;50(5):969-79; discussion 980. doi: 10.1016/j.eururo.2005.12.042. Epub 2006 Jan 30. PMID 16469429
- [Background] Pearce SM, Pariser JJ, Malik RD, Famakinwa OJ, Chung DE. Outcomes following Thulium vapoenucleation of large prostates. Int Braz J Urol. 2016 Jul-Aug;42(4):757-65. doi: 10.1590/S1677-5538.IBJU.2015.0424. PMID 27564287
- [Background] Yu X, Elliott SP, Wilt TJ, McBean AM. Practice patterns in benign prostatic hyperplasia surgical therapy: the dramatic increase in minimally invasive technologies. J Urol. 2008 Jul;180(1):241-5; discussion 245. doi: 10.1016/j.juro.2008.03.039. Epub 2008 May 21. PMID 18499180
- [Background] Elzayat EA, Elhilali MM. Holmium laser enucleation of the prostate (HoLEP): the endourologic alternative to open prostatectomy. Eur Urol. 2006 Jan;49(1):87-91. doi: 10.1016/j.eururo.2005.08.015. Epub 2005 Nov 2. PMID 16314033
- [Background] Kuntz RM, Lehrich K, Ahyai S. Does perioperative outcome of transurethral holmium laser enucleation of the prostate depend on prostate size? J Endourol. 2004 Mar;18(2):183-8. doi: 10.1089/089277904322959842. PMID 15072628
- [Background] Kuntz RM. Current role of lasers in the treatment of benign prostatic hyperplasia (BPH). Eur Urol. 2006 Jun;49(6):961-9. doi: 10.1016/j.eururo.2006.03.028. Epub 2006 Mar 31. PMID 16632179
- See also: www.researchgate.net — https://www.researchgate.net/publication/304340728_Complications_of_Transurethral_Resection_of_the_Prostate
- See also: european association of urology — https://citeseerx.ist.psu.edu/viewdoc/download?doi=10.1.1.601.5664&rep=rep1&type=pdf